CLINICAL TRIAL: NCT00728923
Title: Pilot Study of Minocycline (NPL-2003) in Adults With Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5707
Record Dates: First submitted 2008-07-31; First posted 2008-08-06 (Estimated); Results first posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Minocycline (NPL-2003)
  Interventions: Drug: NPL-2003

INTERVENTIONS:
Drug: NPL-2003 — Minocycline (NPL-2003) daily for 12 weeks
  Other Names: 5707 (Insitution Code name)

SUMMARY:
Obsessive-compulsive disorder (OCD) is a common psychiatric illness that affects up to 2-3% of the population. People with OCD experience anxiety-provoking, intrusive thoughts, known as obsessions, and feel compelled to perform repetitive behaviors, or compulsions. The only medications proven effective for OCD are serotonin reuptake inhibitors (SRIs), but even with SRI treatment, most patients continue to experience significant OCD symptoms, impaired functioning, and diminished quality of life. Recent evidence suggest that a different neurotransmitter, glutamate, may contribute to the symptoms in OCD. Medications that target glutamate hold promise for ameliorating symptoms for those patients continuing to suffer from OCD. In this study we are recruiting patients to receive the drug NPL-2003, which is thought to modulate the neurotransmitter glutamate, added to whatever other OCD medications they are taking in a 12-week open label study.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV Diagnosis of OCD
* Currently on a stable and adequate dose of SRI (or history of prior SRI or CBT treatment meeting criteria for adequate trial)
* Patients not currently receiving an SRI or CBT will be included if they have undergone a prior SRI or CBT trial and they report no interest in pursuing another DRI or CBT trial at this time. Patients who have been on SRIs in the past must be free of SRIs for at least 6 weeks prior to participation
* Y-BOCS score of greater or equal to 16
* Physically health and females must be using effective contraception
* Sufficient severity of symptoms to warrant additional augmentation treatment
* Able to provide consent

Exclusion Criteria:

* Ongoing treatment with other antibiotics and/or Accutane. Patients with lupus erythematosus
* Patients planning to start CBT during the study period or those who have begun CBT within the past 8 weeks
* Presence of psychotic symptoms or lifetime history of schizophrenia, bipolar disorder or other psychotic disorder
* Current major depressive disorder (patients must be free of the disorder for 3 months prior to enrollment). HAM-D must be <18.
* Judged clinically to be at risk of suicide (suicidal ideation, severe depression or other factors
* Current eating disorder
* Severe renal insufficiency
* Documented history of hypersensitivity or intolerance to tetracycline antibiotics
* Concomitant use of anti-coagulant drugs, antacids, iron, calcium, magnesium, aluminum, zinc sales. Note:Concomitant psychotropic medications such as antipsychotics and benzodiazepines will be permitted as long as they have been stable for at least 4 weeks and remain stable during the course of the study.
* Current ETOH/drug abuse or dependence disorder of dependency in the past 3 months
* Female patients who are either pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I. Rodriguez, M.D., Ph.D., Principal Investigator — Columbia-NYSPI-RFMH
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Rodriguez CI, Bender J Jr, Marcus SM, Snape M, Rynn M, Simpson HB. Minocycline augmentation of pharmacotherapy in obsessive-compulsive disorder: an open-label trial. J Clin Psychiatry. 2010 Sep;71(9):1247-9. doi: 10.4088/JCP.09l05805blu. PMID 20923629
- See also: Columbia University Obsessive-Compulsive Disorder Research Clinic — http://www.columbia-ocd.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult outpatients were recruited from the community starting August 2008 until July 2011.
Groups:
- Minocycline: minocycline 100mg bid for 12 weeks
Period: Overall Study
Arm/Group | Minocycline
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Yale-Brown Obsessive-Compulsive Scale
Description: Patients given YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response was defined as at least a 30% reduction on the YBOCS.
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Minocycline: Subjects received minocycline at 50mg BID (twice daily) for 3 days and then at 100mg BID for 12 weeks in addition to their SRI (serotonin reuptake inhibitor).
Arm/Group | Minocycline
Number analyzed (Participants) | 9
participants | 2

2. Secondary Outcome: Number of Patients That Met Response Criteria for the Hamilton Depression Rating Scale.
Description: Patients given HAM-D (Hamilton Depression Scale), a measure of depressive symptoms. For the HAM-D the minimum units are 0 and Maximum units on the total scale are 50. The higher the number on the HAM-D, the more severe the symptoms. Response was defined as at least a 30% reduction on the HAM-D.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Minocycline
Number analyzed (Participants) | 9
participants | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Minocycline
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No